CLINICAL TRIAL: NCT05039853
Title: Improving Mental Health Following Early PREgnancy Loss Using a Brief Cognitive Task
Acronym: IMPREL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21HH6557
Record Dates: First submitted 2021-08-23; First posted 2021-09-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Post-traumatic Stress Disorder; Miscarriage; Ectopic Pregnancy; Pregnancy Loss; Trauma, Psychological
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Abortion, Spontaneous; Pregnancy, Ectopic; Psychological Trauma

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to whether the activity they are assigned to is the experimental intervention or the placebo activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A brief cognitive task-based based intervention (Experimental): Participants will engage in a brief cognitive task including: a memory reminder procedure, playing the computer game, Tetris, on a smart-device using mental rotation +/- Booster.
  Interventions: Behavioral: Brief cognitive task-based intervention
- Placebo activity (Placebo Comparator): Participants will engage with a placebo activity: listening to a pod-cast for approximately 15 minutes on a smart-device.
  Interventions: Behavioral: Placebo activity

INTERVENTIONS:
Behavioral: Brief cognitive task-based intervention — Memory reminder procedure, playing the computer game, Tetris , on a smart-device using mental rotation +/- Boosters
  Arms: A brief cognitive task-based based intervention
Behavioral: Placebo activity — Listening to a pod-cast on a smart-device for approximately 15 minutes.
  Arms: Placebo activity

SUMMARY:
This is a randomised controlled trial designed to investigate the impact of a brief-cognitive task based intervention on intrusive memories, mental health symptoms and daily functioning, in women following an early pregnancy loss.

DETAILED DESCRIPTION:
Women who have experienced an early pregnancy loss (miscarriage or ectopic pregnancy) will be randomly allocated to either a brief cognitive intervention or a placebo activity. Participants will be followed up at week 1, 1 month and 3 months following the intervention. It is hypothesised that those allocated to receive the brief cognitive task-based intervention will develop fever intrusive memories, less severe mental health symptoms and better day to day functioning when compared to women allocated to the placebo activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over
2. Diagnosis of early pregnancy loss (EPL) (missed miscarriage, incomplete miscarriage, complete miscarriage, ectopic pregnancy)
3. Fluent in English
4. Access to a smart device (e.g. phone or tablet)
5. Within 72 hours of EPL (including diagnosis of complete miscarriage or completion of treatment for ectopic pregnancy, missed miscarriage or incomplete miscarriage)

Exclusion Criteria:

1. Women who, in the opinion of the researcher, are unable to give fully informed consent to the study due to for example learning impairment or language barrier.
2. Women with a viable intrauterine pregnancy
3. Women with a pregnancy loss occurring after 20 weeks gestation
4. History of severe mental illness or substance misuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of early pregnancy loss | Week 1
  Number of intrusive memories during the first week following early pregnancy loss recorded by participants in a brief daily diary(morning, afternoon, evening and night) for 7 days.

SECONDARY OUTCOMES:
Number of intrusive memories of early pregnancy loss | Week 5
  Number of intrusive memories during the fifth week following early pregnancy loss recorded by participants in a brief daily diary(morning, afternoon, evening and night) for 7 days.
Character of intrusive memories | Week 1 and week 5
  Character of intrusive memories measured using a numeric scale out of 10 (minimum 1 maximum 10) to rate how vivid and how distressing the intrusive memories were during the first and fifth week following early pregnancy loss
Severity of PTSD symptoms | 1 month and 3 months
  Severity of PTSD measured using the Post-traumatic stress disorder Checklist for DSM-5 (PCL-5) 1 and 3 months following early pregnancy loss. Score range is 0-80 with a higher score representing more severe symptoms.
Frequency and Severity of Functional Impairment | 1 month and 3 months
  Functional impairment measured using the Work and Social Adjustment Scale (WSAS) measured 1 and 3 months following early pregnancy loss. Scores range from 0-40 with the higher score representing worse impairment.
Severity of re-experiencing symptoms cluster | 1 month and 3 months
  Severity of re-experiencing symptoms cluster measured using the re-experincing symptom sub-scale of the Post-traumatic stress disorder Checklist for DSM-5 (PCL-5) at 1 and 3 month following early pregnancy loss. Minimum score 0 maximum score 20 with the higher score being worse.
Number of women meeting the diagnostic threshold for PTSD diagnosis | 1 month and 3 months
  Number of women meeting the diagnostic threshold for PTSD diagnosis measured using the Post-traumatic stress disorder Checklist for DSM-5 (PCL-5) at 1 month and 3 months following early pregnancy loss.
Severity of Anxiety symptoms | 1 month and 3 months
  Severity of anxiety measured using the Hospital Anxiety and Depression Scale (HADS) at 1 and 3 months. Score range 0-21 where 0-7 represents "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe
Severity of Depressions Symptoms | 1 month and 3 months
  Severity of depression measured using the Hospital Anxiety and Depression Scale (HADS) at 1 and 3 months. Score range 0-21 where 0-7 represents "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe.
Number of women meeting the diagnostic threshold for moderate/severe anxiety | 1 month and 3 months
  Number of women meeting the diagnostic threshold for moderate/severe anxiety measured using Hospital Anxiety and Depression Scale (HADS) at 1 and 3 months.Score range 0-21 where 0-7 represents "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe
Number of women meeting the diagnostic threshold for moderate/severe depression | 1 month and 3 months
  Number of women meeting the diagnostic threshold for moderate/severe depression measured using Hospital Anxiety and Depression Scale (HADS) at 1 and 3 months. Score range 0-21 where 0-7 represents "normal," 8-10 "mild," 11-14 "moderate," and 15-21 "severe

OTHER OUTCOMES:
The relationship between number of intrusive memories of early pregnancy loss and 1. Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | Week 1 , week 5, 1 month and 3 months
  The relationship between the number of intrusive memories of early pregnancy loss and 1. Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.
The relationship between the severity of PTSD symptoms and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | 1 month and 3 months
  The relationship between the severity of PTSD symptoms measured at 1 and 3 months and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.
The relationship between the number of women who reach PTSD diagnostic thresholds and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | 1 and 3 months
  The relationship between the number of women who reach PTSD diagnostic threshold at 1 and 3 months and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.
The relationship between the severity of functional impairment measured at 1 and 3 months and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | 1 and 3 months
  The relationship between the severity of functional impairment measured at 1 and 3 months and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.
The relationship between the severity of symptoms of anxiety and depression, and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | 1 and 3 months
  The relationship between the severity of symptoms of anxiety and depression, and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.
The relationship between the number of women who meet anxiety or depression diagnostic thresholds and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy. | 1 and 3 months
  The relationship between the number of women who meet diagnostic thresholds for moderate/severe anxiety or depression and 1.Type of early pregnancy loss and management 2. Timing of traumatic event 3. Recurrent early pregnancy loss 4. Ethnicity and 5. Subsequent pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bourne, Principal Investigator — Imperial College London
Locations (1):
- Imperial college healthcare NHS trust, London, United Kingdom